CLINICAL TRIAL: NCT04379193
Title: Ambulatory Neuroproprioceptive Facilitation and Inhibition Physical Therapy Does Not Modulate Serum Level of Neuroactive Steroids
Brief Title: Physical Therapy and Neuroactive Steroids Therapy Does Not Modulate Serum Level of Neuroactive Steroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VP/22/0/2014/1
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
Keywords: neuroactive steroids; physical therapy; dehydroepiandrosterone; cortisol; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor program activating therapy (Experimental): MPAT is method developed and verified by our team. In this therapy, patients are corrected into a postural position where the joints are functionally centered. Somatosensory (manual and verbal) stimuli are then applied to activate motor programs in the brain, which then lead to the co-contraction of the patient's whole body when laying, sitting, standing up or moving forward. Activated programs are repeated under various conditions and in different situations and environments to teach the patients to automatically use the acquired motor skills in daily life. Therapy was realized within the ambulatory area of the Department of Neurology at Kralovske Vinohrady University Hospital in Prague.
  Interventions: Behavioral: Neuroproprioceptive facilitation and inhibition physical therapy
- Vojta's reflex locomotion (Experimental): VRL is a standard approach for patients with MS in the Czech Republic. In the therapy, global patterns of the reflex locomotion are activated by stimulation of specific zones, with the individual placed in a precisely determined initial position (supine, prone and side laying, low kneeling position). These movement patterns have the qualities of the forward movement (locomotion) and the movement responses are precisely defined. Reflex locomotion (reflex turning and reflex creeping) is used in therapy to activate involuntarily responses of muscle function, which are necessary for spontaneous movements. Therapy was realized at the Department of Rehabilitation and Sport Medicine at Motol University Hospital.
  Interventions: Behavioral: Neuroproprioceptive facilitation and inhibition physical therapy

INTERVENTIONS:
Behavioral: Neuroproprioceptive facilitation and inhibition physical therapy — All groups underwent two months' therapy, 16 face-to-face sessions (1 hour, twice a week for two months).

SUMMARY:
This study describes modulation of neuroproprioceptive facilitation and inhibition physical therapy on serum level of neuroactive steroids in multiple sclerosis.

DETAILED DESCRIPTION:
In the parallel group, single blind, randomized controlled trial, participant underwent two kinds of neuroproprioceptive PT (MPAT and VRL). At baseline and after the end of the two months' therapeutic program, a blinded assessor evaluated clinical outcomes and data from serum level.

ELIGIBILITY:
Inclusion Criteria:

* prevailed spastic paraparesis, stable clinical status and treatment in the preceding 3 months determined by neurologist,
* Expanded Disability Status Scale score (EDSS) max. 7.5

Exclusion Criteria:

* other neurological disease or conditions disabling movement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
serum level of neuroactive steroids | 2 months
  cortisol, cortisone, 7 alfa-OH-DHEA, 7 beta-OH-DHEA, 7 oxo- oxo-DHEA, DHEA

SECONDARY OUTCOMES:
Berg Balance Scale, BBS outcomes | 2 months
  14 items objective measure of static balance and risk of falls (0 the best, 56 the worse)
Paced Auditory Serial Addition Test | 2 months
  The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it.
the 29-item Multiple Sclerosis Impact Scale, MSIS -29 | 2 months
  a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
Modified Fatigue Impact Scale | 2 months
  The MFIS is generally presented as a 21-item questionnaire, but there's also a 5-question version. Most people fill it out on their own in a doctor's office. Expect to spend anywhere from five to ten minutes circling your answers.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, Ph.D., Principal Investigator — Third Faculty of Mecicine, Charles Univerzity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angelova G, Skodova T, Prokopiusova T, Markova M, Hruskova N, Prochazkova M, Pavlikova M, Spanhelova S, Stetkarova I, Bicikova M, Kolatorova L, Rasova K. Ambulatory Neuroproprioceptive Facilitation and Inhibition Physical Therapy Improves Clinical Outcomes in Multiple Sclerosis and Modulates Serum Level of Neuroactive Steroids: A Two-Arm Parallel-Group Exploratory Trial. Life (Basel). 2020 Oct 31;10(11):267. doi: 10.3390/life10110267. PMID 33142850